CLINICAL TRIAL: NCT02694419
Title: Effect of Body Weight on Endometrial Ultrasonographic Characteristics in Polycystic Ovary Syndrome Patients
Brief Title: The Effect of Obesity on Endometrium in PCOS
Acronym: OB-PCO
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Mohamed Abbas, Dr, Assiut University
Other Study IDs: PCOS
Record Dates: First submitted 2016-02-24; First posted 2016-02-29 (Estimated); Last update posted 2017-08-11 (Actual); Status verified 2017-08

CONDITIONS: Body Weight; Polycystic Ovary Syndrome
Keywords: endometrium
MeSH Terms: conditions — Body Weight; Polycystic Ovary Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- obese/PCO: Women with PCOS who are overweight\obese with BMI ≥ 25 kg/m2.
  Interventions: Device: Doppler evaluation
- normal weight/PCO: Women with PCOS who are normal weight with BMI < 25 kg/m2.
  Interventions: Device: Doppler evaluation
- Obese/fertile: Fertile regularly menstruating women with at least one previous spontaneous pregnancy who are overweight\obese with BMI ≥ 25 kg/m2.
  Interventions: Device: Doppler evaluation
- normal weight/fertile: Fertile regularly menstruating women with at least one previous spontaneous pregnancy who are normal weight with BMI < 25 kg/m2.
  Interventions: Device: Doppler evaluation

INTERVENTIONS:
Device: Doppler evaluation — Endometrial volume, endometrial and subendometrial vascularity indices are measured by 3D power Doppler

SUMMARY:
The effect of Polycystic Ovary Syndrome (PCOS) with or without obesity has received a few attentions. There is a lack of evidence to whether the BMI affects the endometrial blood flow, which is necessary for implantation.

ELIGIBILITY:
Inclusion Criteria:

* Women with PCOS are diagnosed according to Rotterdam criteria, (Rotterdam and ASRM-Sponsored, 2004)by the presence of two out of the following three: oligomenorrhea (absence of menses for 35-182 days) or amenorrhea (absence of menses for >182 days), signs or symptoms of hyperandrogenism (acne, hirsutism), US showing polycystic ovaries.
* Fertile women had regular menstruation, with at least one previous spontaneous pregnancy.

Exclusion Criteria:

* Women known to have hepatic or renal dysfunction, Diabetes mellitus, hypertension, or cardiovascular disease.
* If they have used induction of ovulation drugs for the last three months.
* If they have used hormonal contraception in the last three months.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: 100 women were recruited from gynecology clinic of Women Health Hospital
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
the mean difference in Doppler indices (VI-FI-VFI) | 24 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Ahmed Abbas, Assiut, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No